CLINICAL TRIAL: NCT02370641
Title: Variations in Urolithin Production by the Microbiome After Pomegranate Extract Administration: Understanding Metabolism and Responsiveness to Pomegranate Ellagitannins
Brief Title: Effects of Pomegranate Extract on Intestinal Flora
Acronym: PomX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 12-000874
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Urolith
Keywords: urolithin A; microflora
MeSH Terms: conditions — Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- urolithin excretors (Active Comparator): The excretor status will be determined by analysis for urolithin A glucuronide in 24 hour urine after one dose of POMx. A blood sample and stool sample will be obtained before administering the extract.
  Interventions: Dietary Supplement: PomX
- non excretors (Active Comparator): The excretor status will be determined by analysis for urolithin A glucuronide in 24 hour urine after one dose of POMx. A blood sample and stool sample will be obtained before administering the extract.
  Interventions: Dietary Supplement: PomX

INTERVENTIONS:
Dietary Supplement: PomX — 1000 mg POMx daily for 4 weeks

SUMMARY:
A total of 20 individuals, 10 urolithin excretors and 10 nonexcretors will be enrolled. The excretor status will be determined by analysis for urolithin A glucuronide in 24 hour urine after one dose of POMx. A blood sample and stool sample will be obtained before administering the extract. Subjects will be asked to consume one capsule of 1000 mg POMx daily for 4 weeks. At day 28, a blood sample, 24 hour urine sample will be obtained, and the stool collected by the participant in the prior 24 hours will be returned to the Center. Blood and urine urolithin, ellagic acid levels and stool bacteria enumeration and identification (including pyrosequencing) will be measured with the samples collected. A stool DNA sample will be preserved and frozen for potential future measurement of gene-nutrient interaction in pomegranate metabolism.

Throughout the study participants will be instructed not to consume pomegranate products, walnuts, or polyphenol-rich fruits ((strawberry, raspberry etc) or juices drawn from a list used in prior studies. The study will be carried out in accordance with the guidelines of the Human Subjects Protection Committee of the University of California, Los Angeles. All subjects will give written informed consent before the study begins. Participants will be recruited by advertisement in the local newspaper in the Los Angeles Area close to UCLA.

DETAILED DESCRIPTION:
At screening, informed consent and health insurance portability and assurance (HIPAA) authorization will be reviewed and signed. A medical history will be obtained. If criteria for enrollment are satisfied, a fasting blood sample will be collected for a comprehensive metabolic panel, and blood count. Results will be reviewed by the study physician for compliance to inclusion and exclusion criteria. The screening visit will also include a review of foods to avoid during run-in and study participation. Once lab results from the screening visit come back and are determined to be satisfactory for inclusion, the subject will be called and instructed to start dietary restrictions. The first stool collection (Day -1) will occur after two weeks of dietary compliance.

Day -1: Subjects will be asked to collect an entire stool and store it in a cooler filled with ice packs, along with a collection container until delivery to the lab within 24 hours.

Day 1: Subjects will take the 1st dose of POMx and be given a container for collecting their urine for 24 hours and asked to refrigerate this as the urine is collected. This urine will be used to determine the presence of urolithin A and whether they are "responder or non responder". Participants will be asked to consume 1 POMx capsule daily and to abstain from consuming pomegranates, walnuts, or polyphenol-rich foods or juices drawn from a list.

Day 27: Subjects will collect one entire stool and place in the provided cooler filled with ice packs for storage of the stool sample until delivery to the lab within 24 h. Urine collection will start at 8am after the morning dose of POMx and last until 8 am the day of clinic visit.

Day 28: Stool and urine sample will be collected. The stool sample collected at home (within the prior 24 hours) will be returned on this day. Blood sample will be collected. Compliance will be assessed by pill count. Safety and tolerance data will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-50 years of age at screen.
2. In good health
3. Subjects must read and sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or enrollment. A subject will be excluded for any condition that might compromise the ability to give truly informed consent.

Exclusion Criteria:

1. Any history of gastrointestinal disease except for appendectomy
2. Any use of antibiotics or laxatives during the 2 months prior to study enrollment.
3. Any subject with a history of diabetes mellitus, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP>160mmHg, diastolic BP>95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history or routine physical examination.
4. Any subject consuming pre- or probiotics
5. Any subject with a screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator.
6. Any subject who currently uses tobacco products or has used tobacco products within the last year.
7. Any subject who is unable or unwilling to comply with the study protocol.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, M.D., Ph.D., Principal Investigator — UCLA Department of Medicine, Division of Clinical Nutrition

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD with other researchers.

REFERENCES:
- [Result] Li Z, Henning SM, Lee RP, Lu QY, Summanen PH, Thames G, Corbett K, Downes J, Tseng CH, Finegold SM, Heber D. Pomegranate extract induces ellagitannin metabolite formation and changes stool microbiota in healthy volunteers. Food Funct. 2015 Aug;6(8):2487-95. doi: 10.1039/c5fo00669d. Epub 2015 Jul 20. PMID 26189645

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period was 10/31/2012 - 7/2/2013. Enrollment took place in a private setting in the clinic located at the site.
Pre-assignment Details: Twenty-six healthy participants were enrolled in the study. There were two study phases including a 2-week run-in period and a 4-week intervention period. Six subjects who did not complete the study were excluded.
Groups:
- Urolithin Excretors: The excretor status was determined by analysis of urolithin A glucuronide in 24 hour urine after one dose of POMx. A blood sample and stool sample were obtained before administering the extract.
  PomX: 1000 mg POMx daily for 4 weeks
- Non Excretors: The excretor status was determined by the analysis of urolithin A glucuronide in 24 hour urine after one dose of POMx. A blood sample and stool sample were obtained before administering the extract.
  PomX: 1000 mg POMx daily for 4 weeks
Period: Overall Study
Arm/Group | Urolithin Excretors | Non Excretors
Started | 18 | 8
Completed | 14 | 6
Not Completed | 4 | 2
Not completed — dropped study | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Urolithin Excretors | Non Excretors | Total
Number analyzed (Participants) | 14 | 6 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 6 | 20
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 8 | 3 | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 12 | 2 | 14
  Black | 0 | 2 | 2
  Asian | 2 | 2 | 4
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23 (3) | 23 (3) | 23 (3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Total Microflora Between Urolithin Excretors and Non-excretors
Description: Difference of percentage of total microflora between urolithin excretors and non-excretors after consumption of pomegranate extract for 4 weeks
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: percentage of total microflora
Groups:
- Microbial Phylum Abundance in Urolithin Excretors; Microbial Phylum Abundance in Non Excretors: Microbial phylum abundance (% of total) in urolithin excretors after consumption of 1000 mg pomegranate extract daily for 4 weeks
Arm/Group | Microbial Phylum Abundance in Urolithin Excretors | Microbial Phylum Abundance in Non Excretors
Number analyzed (Participants) | 14 | 6
percentage of total microflora
  Percentage of phylum Firmecutes at baseline | 60 (10.1) | 68 (17.2)
  Percentage of phylum Firmecutes at week 4 | 56 (10.5) | 70 (9.3)
  Percentage of phylum Proteobacteria at baseline | 3.4 (2.5) | 2.5 (1.4)
  Percentage of phylum Proteobacteria at week 4 | 6 (5.4) | 1.8 (0.5)
Statistical Analysis 1: Comparison: Microbial Phylum Abundance in Urolithin Excretors vs Microbial Phylum Abundance in Non Excretors; Comparison was made to week 4 minus baseline change of phylum Firmicutes abundance between urolithin excretors and non excretors; Test type: Other; p = 0.012, Wilcoxon (Mann-Whitney) — p<0.05 is defined as significant; Mean Difference (Final Values) = -4
Statistical Analysis 2: Comparison: Microbial Phylum Abundance in Urolithin Excretors vs Microbial Phylum Abundance in Non Excretors; Comparison was made to week 4 minus baseline change of phylum Proteobacteria abundance between urolithin excretors and non excretors; Test type: Other; p = 0.009, Wilcoxon (Mann-Whitney) — p<0.05 was defined as significant; Mean Difference (Final Values) = 2.6

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 4 week period
Description: Participants were monitored and questioned regarding the occurrence and nature of any adverse experiences.
Groups:
- Microbial Phylum Abundance in Urolithin Excretors: microbial phylum abundance in urolithin excretors after consumption of 1000 mg pomegranate extract daily for 4 weeks
- Microbial Phylum Abundance in Urolithin Non Excretors: The excretor status was determined by the analysis of urolithin A glucuronide in 24 hour urine after one dose of POMx. A blood sample and stool sample were obtained before administering the extract.
  PomX: 1000 mg POMx daily for 4 weeks
Arm/Group | Microbial Phylum Abundance in Urolithin Excretors | Microbial Phylum Abundance in Urolithin Non Excretors
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/6
Other Adverse Events (participants affected / at risk) | 2/14 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microbial Phylum Abundance in Urolithin Excretors (N=14) | Microbial Phylum Abundance in Urolithin Non Excretors (N=6)
nausea after taking supplement on empty stomach (Gastrointestinal disorders) | 1 (1) | 1 (1)
mild gastrointestinal discomfort after taking supplement on empty stomach (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No